CLINICAL TRIAL: NCT01703078
Title: A Phase 1 Exploratory Trial Evaluating Safety and Tolerability of Topical Administration of Different Concentrations of an Ingenol Derivative Compared to Ingenol Mebutate Gel 0.05% Applied on Two Consecutive Days to Four Separate 25cm2 Treatment Areas on the Forearms of Subjects With Actinic Keratosis (Field Therapy)
Brief Title: Safety and Tolerability of Different Concentrations of an Ingenol Derivative Field Therapy in the Treatment of Actinic Keratosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: LP0084-68
Record Dates: First submitted 2012-10-05; First posted 2012-10-10 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2013-02

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ingenol mebutate gel 0.05% (Active Comparator): once daily for two consecutive days
  Interventions: Drug: Ingenol once daily for two consecutive days
- Ingenol derivative concentration 1 (Experimental): once daily for two consecutive days
  Interventions: Drug: Ingenol once daily for two consecutive days
- Ingenol derivative concentration 2 (Experimental): once daily for two consecutive days
  Interventions: Drug: Ingenol once daily for two consecutive days
- Ingenol derivative concentration 3 (Experimental): once daily for two consecutive days
  Interventions: Drug: Ingenol once daily for two consecutive days

INTERVENTIONS:
Drug: Ingenol once daily for two consecutive days

SUMMARY:
The purpose of this study is to determine if the new ingenol derivative gels are as safe as and as well tolerated as ingenol mebutate gel when applied to AK lesions on the forearm for two consecutive days.

DETAILED DESCRIPTION:
Various concentrations of new ingenol derivatives will be applied to AKs on the forearms. Reactions and safety will be compared to a US registered and marketed ingenol gel to ascertain if the new ingenol is at least as safe and as well tolerated as the registered ingenol.

ELIGIBILITY:
Inclusion Criteria:

* Must be male or female and at least 18 years of age.
* Female patients must be of non-childbearing potential or if of childbearing potential then negative serum and urine pregnancy test and using effective contraception
* Ability to provide informed consent

Exclusion Criteria:

* location of the selected treatment area within 5cm of an incompletely healed wound or within 5cm of a suspected basal cell carcinoma or squamous cell carcinoma
* undergone Cosmetic or therapeutic procedures within 2cm of the selected treatment area in the 2 weeks prior to Visit 2
* use of acid-containing therapeutic products within 2cm of the selected treatment area in the 2 weeks prior to Visit 2
* use of topical moisturisers/creams/lotions, artificial tanners or topical steroids within 2cm of the selected treatment areas in the 2 weeks prior to visit 2 Treatment with immunomodulators, or interferon/interferon inducers or systemic medications that suppress the immune system within 4 weeks of Visit 2
* Treatment with 5-FU, imiquimod, diclofenac, or photodynamic therapy within 2 cm of the treatment area in the 8 weeks prior to visit 2
* use of systemic retinoids
* those who are currently participating in any other clinical trial
* females who are pregnant or are breastfeeding
* those known or suspected of not being able to comply with the requirements of the protocol or provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Safety of a new ingenol derivative compared to ingenol mebutate gel applied topically once daily for two consecutive days to four separate treatment areas containing actinic keratosis on the forearm | 8 weeks
  Safety data to be collected via CRF entries of AEs/SAEs and photographs.

SECONDARY OUTCOMES:
Evaluate treatment responses on Actinic Keratosis of different concentrations of a new ingenol derivative gel compared to the ingenol mebutate gel as assessed by reduction in number of clinically visible selected AK lesions eight weeks after treatment | 8 weeks
  Assessed by Reflective Confocal Microscopy scoring of visible selected AK lesions

CONTACTS AND LOCATIONS:
Overall Officials: Hans P Soyer, Principal Investigator — Dermatology Department, Brisbane Public Hospital
Locations (1):
- Dermatology Department, Woolloongabba, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: LEO Pharma — http://www.leopharma.com
- See also: Therapeutic Goods Administration — http://www.tga.gov.au